CLINICAL TRIAL: NCT02819752
Title: Phase I Dose-escalation Study of PEmbrolizumab (MK3475) Anti-PD1 Immune Checkpoint Inhibitor Combined With Radical Chemoradiotherapy in Patients With Stage IV Squamous Cell Carcinoma of the Head and Neck
Brief Title: PEmbrolizumab Combined With Chemoradiotherapy in Squamous Cell Carcinoma of the Head and Neck
Acronym: PEACH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: funding pulled
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCR4325
Record Dates: First submitted 2016-06-22; First posted 2016-06-30 (Estimated); Results first posted 2025-12-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinoma
Keywords: squamous cell carcinoma; squamous cell carcinoma of the head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — pembrolizumab; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HPV-ve stage IVA/IVB SCCHN (Experimental): Pembrolizumab and Chemoradiotherapy
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy; Drug: Chemotherapy
- HPV+ve stage IVA/IVB SCCHN (Experimental): Pembrolizumab and Chemoradiotherapy
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab
  Other Names: MK-3475/pembrolizumab (KEYTRUDA®)
Radiation: Radiotherapy — Radiotherapy - Standard Treatment
Drug: Chemotherapy — Chemotherapy - Standard Treatment

SUMMARY:
This study aims to establish whether the combination of pembrolizumab (MK-3475) and conventional cisplatin-based chemoradiotherapy is tolerable and results in acceptable levels of acute and late toxicity in patients with stage IV LA-SCCHN. In particular, the study will provide data on the levels of mucosal and cutaneous toxicity within the radiation fields, as these are the primary acute toxicities associated with this treatment regimen. In addition, toxicity outside the radiation portals (which may theoretically be exacerbated by radiation) will be studied. However, all toxicity will be monitored. This study will also give an indication of the activity of pembrolizumab in LA-SCCHN because we are deliberately selecting a group of patients with high- and intermediate-risk disease who have a significant chance of experiencing loco-regional or systemic failure.

DETAILED DESCRIPTION:
This will be a single centre phase 1 dose-escalation study to confirm the safety of combining pembrolizumab with standard platin-based chemoradiotherapy in patients with stage IV high- and intermediate-risk locally-advanced squamous cell carcinoma of the head and neck (LA-SCCHN). 6-36 patients (18 HPV+ve and 18 HPV-ve) will be recruited in a standard 3+3 dose-escalation trial design with an expansion cohort at the maximum tolerated dose (or 200 mg, if no DLT is defined). A pre-loading dose of 100 or 200mg (dependent on dosing level) of pembrolizumab will be given once the patient has completed the screening period. Patients will then return 2 weeks later to begin cycle 1 of a regimen of pembrolizumab 3 weekly at a dose of 100 or 200mg (dependent on dosing level) for a total of 7 cycles (3 during chemoradiotherapy and 4 after chemoradiotherapy).

Parallel studies in HPV-ve and HPV +ve disease will be conducted (note these patients may have different patterns of co-morbidity and, hence, different treatment-related toxicities). The primary endpoint of the study will be safety and tolerability. Dose-limiting acute toxicity will be assessed during administration of study drug according to CTCAEv4.0. The maximum tolerated dose of study drug (or 200 mg in the absence of DLT) will be used in a subsequent randomised phase 2 study comparing standard-of-care therapy with standard-of-care therapy plus study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Have treatment naive and histologically confirmed high-/intermediate-risk LA-SCCHN
2. Be willing and able to provide written informed consent for the trial.
3. Be > or = 18 years of age on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1.
5. Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumour lesion.
6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
7. Be fit for definitive platin-based chemoradiation therapy.
8. Demonstrate adequate organ function as defined in table 1, all screening labs should be performed within 10 days of confirmation of study eligibility.
9. Female patient of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to confirmation of study eligibility. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female patient s of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 6.7.2). Patient s of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male patient s should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has received prior radiotherapy to the head and neck region.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has had a prior monoclonal antibody, chemotherapy, targeted small molecule therapy, or radiation therapy.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patient s with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
7. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Patient s with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patient s with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has active tuberculosis.
11. Has known hypersensitivity to pembrolizumab or any of its excipients.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Kevin Harrington, CTU, Study Director — Consultant Clinical Oncologist
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the period between July 2017 and July 2019, 3 patients were recruited to the study at the Royal Marsden Hospital in the United Kingdom.
Groups:
- HPV-ve Stage IVA/IVB SCCHN; HPV+ve Stage IVA/IVB SCCHN: Pembrolizumab and Chemoradiotherapy
  Pembrolizumab: Pembrolizumab administered as a 30-minute infusion. Dose level 1: 100mg 3-weekly; dose level 2: 200mg 3-weekly.
  Radiotherapy: Radiotherapy - Standard Treatment
  Chemotherapy: Chemotherapy - Standard Treatment
Period: Overall Study
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Started | 0 | 3
Completed | 0 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients consented and registered to participate in the trial constitute baseline analysis population. Three patients were recruited to HPV+ve arm and no patients were recruited to HPV-ve arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN | Total
Number analyzed (Participants) | 0 | 3 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 2 | 2
  >=65 years |  | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 3 | 3
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom |  | 3 | 3
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants]
  0 = Normal activity. |  | 1 | 1
  1 = Symptoms, but ambulatory. |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Patients With Dose Limiting Toxicities (DLT).
Description: To establish the maximum tolerated dose that can safely be combined with platin-based chemoradiotherapy in patients with HPV-ve and HPV+ve LA-SCCHN.
Time Frame: Six weeks after the completion of chemoradiotherapy
Population: All patients registered on the trial and have received at least one treatment dose. Only three patients were treated with one of the doses and the trial terminated early. Maximum Tolerated Dose was not established.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Number analyzed (Participants) | 0 | 3
Participants |  | 0

2. Primary Outcome: Acute Toxicity as Measured During Treatment by CTCAE v4.0
Description: Count and percentage of patients with any CTCAE graded toxicity from start of trial treatment until 6 weeks following end of treatment
Time Frame: Up until 6 weeks after the end of chemoradiotherapy (week 14 of the study)
Population: All patients registered on the trial and have received at least one treatment dose.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Number analyzed (Participants) | 0 | 3
Participants
  Number of patients with any grade 1 or more toxicities |  | 3
  Number of patients with any grade 2 or more toxicities |  | 3

3. Secondary Outcome: Percentage of Progression Free Survival at 6, 12 and 24 Months Post Treatment Start.
Description: Calculated as percentage of evaluable patients alive and disease free at each time point.
Time Frame: Six months, one year and two years
Population: All patients registered on the trial and have received at least one treatment dose.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Number analyzed (Participants) | 0 | 3
Participants
  Number of patients progression free at 6 months |  | 3
  Number of patient progression free at 12 months |  | 3
  Number of patients progression free at 24 months: number analyzed (Participants) | 0 | 1
  Number of patients progression free at 24 months |  | 1

4. Secondary Outcome: Percentage of Overall Survival at 6, 12 and 24 Months
Description: Calculated as percentage of evaluable patients alive at each time point
Time Frame: Six months, one year and two years
Population: All patients registered on the trial and have received at least one treatment dose.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Number analyzed (Participants) | 0 | 3
Participants
  Number of patients alive at 6 months |  | 3
  Number of patients alive at 12 months |  | 3
  Number of patients alive at 24 months: number analyzed (Participants) | 0 | 1
  Number of patients alive at 24 months |  | 1

5. Secondary Outcome: Percentage of Patients With Clinical Benefit (CR/PR/SD) Using RECIST at 6, 12 and 24 Months
Description: Calculated as percentage of evaluable patients with clinical benefit (CR/PR/SD) using RECIST at 6, 12 and 24 months
Time Frame: Six months, one year and two years
Population: All patients who consented and received trial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Number analyzed (Participants) | 0 | 3
Participants
  Number of patients with CR/PR/SD response at 6 months |  | 3
  Number of patients with CR/PR/SD response at 12 months |  | 3
  Number of patients with CR/PR/SD response at 24 months: number analyzed (Participants) | 0 | 1
  Number of patients with CR/PR/SD response at 24 months |  | 1

6. Secondary Outcome: Percentage of Patients With Any Grade 1 Plus RTOG Toxicities
Description: Calculated as percentage of patients with any grade 1 toxicities from start of treatment up to 52 weeks from the end of radiotherapy.
Time Frame: 52 weeks from the end of radiation therapy (week 7)
Population: Patients who consented and received the combination therapy
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Number analyzed (Participants) | 0 | 3
Participants |  | 3

7. Other Pre Specified Outcome: Identify Biomarkers and Correlate With Clinical Benefit, as Defined by RECIST v1.1
Description: Mean biomarker levels in patients according to the categories of RECIST response CR/PR/SD vs PD).
Time Frame: through study completion (24 months)
Population: All patients who consented and received trial treatment. Data not available for this outcome, the planned laboratory work was not performed as the smaller than planned sample size meant this was not thought to be useful.
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Analysis of Circulating Free Tumour DNA
Description: Description of circulating free tumour DNA levels by time to progression.
Time Frame: Screening, week 3, week 9 and week 15
Population: as for outcome 7
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Immunohistochemical Analysis to Identify Immune Infiltrates
Description: Description of laboratory findings from the immunohistochemical analysis of tissue samples.
Time Frame: through study completion (24 months)
Population: as for outcome 7
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the first dose of pembrolizumab until the patients 12 weeks safety follow-up visit.
Description: No patients were recruited to HPV-ve arm, therefore no adverse events were reported for this arm.
Arm/Group | HPV-ve Stage IVA/IVB SCCHN | HPV+ve Stage IVA/IVB SCCHN
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/3
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPV-ve Stage IVA/IVB SCCHN (N=0) | HPV+ve Stage IVA/IVB SCCHN (N=3)
Febrile Neutropenia (Blood and lymphatic system disorders) | NA | 1 (1)
Vomiting (Gastrointestinal disorders) | NA | 1 (1)
Nausea (Gastrointestinal disorders) | NA | 1 (1)
Fever (General disorders) | NA | 2 (4)
Anorexia (Metabolism and nutrition disorders) | NA | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPV-ve Stage IVA/IVB SCCHN (N=0) | HPV+ve Stage IVA/IVB SCCHN (N=3)
Anemia (Blood and lymphatic system disorders) | NA | 1 (5)
Tinnitus (Ear and labyrinth disorders) | NA | 3 (7)
Ear Pain (Ear and labyrinth disorders) | NA | 1 (1)
Hearing Impaired (Ear and labyrinth disorders) | NA | 1 (1)
Other (Ear and labyrinth disorders) | NA | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | NA | 3 (6)
Dry Mouth (Gastrointestinal disorders) | NA | 3 (8)
Oral Pain (Gastrointestinal disorders) | NA | 2 (3)
Constipation (Gastrointestinal disorders) | NA | 2 (3)
Dysphagia (Gastrointestinal disorders) | NA | 2 (2)
Diarrhea (Gastrointestinal disorders) | NA | 1 (1)
Stomach Pain (Gastrointestinal disorders) | NA | 1 (1)
Gastritis (Gastrointestinal disorders) | NA | 1 (1)
Dyspepsia (Gastrointestinal disorders) | NA | 1 (1)
Other (Gastrointestinal disorders) | NA | 2 (3)
Vomiting (Gastrointestinal disorders) | NA | 1 (1)
Nausea (Gastrointestinal disorders) | NA | 2 (2)
Flu Like Symptoms (General disorders) | NA | 1 (1)
Fatigue (General disorders) | NA | 1 (1)
Neck Edema (General disorders) | NA | 1 (1)
Other (General disorders) | NA | 1 (1)
Upper Respiratory Infection (Infections and infestations) | NA | 1 (1)
Other (Infections and infestations) | NA | 1 (1)
Dermatitis Radiation (Injury, poisoning and procedural complications) | NA | 3 (5)
Neutrophil Count Decreased (Investigations) | NA | 1 (2)
Platelet Count Decreased (Investigations) | NA | 1 (2)
Blood Bilirubin Increased (Investigations) | NA | 1 (1)
Alanine Aminotransferase Increased (Investigations) | NA | 2 (5)
Aspartate Aminotransferase Increased (Investigations) | NA | 2 (3)
GGT Increased (Investigations) | NA | 2 (6)
Alkaline Phosphatase (Investigations) | NA | 2 (2)
Weight Loss (Investigations) | NA | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | NA | 1 (2)
Dehydration (Metabolism and nutrition disorders) | NA | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | NA | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | NA | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | NA | 2 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | NA | 1 (1)
Dysgeusia (Nervous system disorders) | NA | 2 (4)
Headache (Nervous system disorders) | NA | 2 (2)
Myelitis (Nervous system disorders) | NA | 1 (1)
Other (Nervous system disorders) | NA | 1 (1)
Insomnia (Psychiatric disorders) | NA | 3 (3)
Anxiety (Psychiatric disorders) | NA | 2 (2)
Suicidal Ideation (Psychiatric disorders) | NA | 1 (1)
Premature Menopause (Reproductive system and breast disorders) | NA | 1 (1)
Vaginal Dryness (Reproductive system and breast disorders) | NA | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | NA | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | NA | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | NA | 2 (2)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | 2 (2)
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Other (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | NA | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | NA | 2 (3)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | NA | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | NA | 1 (1)
Other (Skin and subcutaneous tissue disorders) | NA | 1 (1)
Lymphedema (Vascular disorders) | NA | 1 (1)
Bruising (Injury, poisoning and procedural complications) | NA | 1 (1)
Hypothyroidism (Endocrine disorders) | NA | 1 (1)
Fever (General disorders) | NA | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT02819752/Prot_SAP_000.pdf